CLINICAL TRIAL: NCT04682379
Title: The Role of Proprioceptive Deficits in the Progression of Adolescent Idiopathic Scoliosis
Brief Title: Adolescent Idiopathic Scoliosis and Proprioceptive Defect
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 20-525
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-01

CONDITIONS: Adolescent Idiopathic Scoliosis; Idiopathic Scoliosis; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoliotic patients with proprioceptive deficits: Study subjects possessed statistically significant differences in testing outcomes of proprioception compared with healthy controls.
  Interventions: Diagnostic Test: Proprioceptive assessment
- Scoliotic patients without proprioceptive deficits: Study subjects with similar testing results of proprioception compared with healthy controls.
  Interventions: Diagnostic Test: Proprioceptive assessment

INTERVENTIONS:
Diagnostic Test: Proprioceptive assessment — 1. Trunk flexion-extension repositioning test
  2. Trunk lateral-flexion repositioning test
  3. Trunk axial-rotation repositioning test
  4. Neck rotation repositioning test
  5. Elbow flexion repositioning test
  6. Knee extension repositioning test

SUMMARY:
This is the first clinical study to examine the spinal and peripheral proprioceptive deficits in longitudinal terms among subjects with adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of adolescent idiopathic scoliosis
* did not receive or failed conservative treatment

Exclusion Criteria:

* spinal injury, fracture, or spinal tumour
* neurological deficit
* brain or spinal cord abnormality
* developmental delay
* psychological disorder

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Potential participants will be identified by consecutively screening in the clinics of the speciality outpatient department at the Hospital for all patients with scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Repositioning errors | Baseline
  The deviation between the position achieved by the subject and the reference position.
Repositioning errors | One year follow-up
  The deviation between the position achieved by the subject and the reference position.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cheung, Principal Investigator — The University of Hong Kong
Locations (1):
- The Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lau KKL, Law KKP, Kwan KYH, Cheung JPY, Cheung KMC, Wong AYL. Timely Revisit of Proprioceptive Deficits in Adolescent Idiopathic Scoliosis: A Systematic Review and Meta-Analysis. Global Spine J. 2022 Oct;12(8):1852-1861. doi: 10.1177/21925682211066824. Epub 2021 Dec 15. PMID 34911378
- [Background] Lau KKL, Law KKP, Kwan KYH, Cheung JPY, Cheung KMC. Proprioception-related gene mutations in relation to the aetiopathogenesis of idiopathic scoliosis: A scoping review. J Orthop Res. 2023 Dec;41(12):2694-2702. doi: 10.1002/jor.25626. Epub 2023 Jun 4. PMID 37203456
- [Background] Lau KK, Kwan KY, Cheung JP, Chow W, Law KK, Wong AY, Chow DH, Cheung KM. Reliability of a three-dimensional spinal proprioception assessment for patients with adolescent idiopathic scoliosis. Eur Spine J. 2022 Nov;31(11):3013-3019. doi: 10.1007/s00586-022-07338-0. Epub 2022 Aug 3. PMID 35922635